CLINICAL TRIAL: NCT05639504
Title: Sepsis Prognosis and Diagnosis in the Emergency Department Using a Host Response Classifier (SPEED) UK - a Multi-Centre Observational Study
Brief Title: Sepsis Prognosis and Diagnosis in the Emergency Department (SPEED)
Status: Withdrawn | Type: Observational
Why Stopped: Study never started, change in company focus on US
Sponsor: Inflammatix (Industry)
Responsible Party: Sponsor
Other Study IDs: INF-25
Record Dates: First submitted 2022-09-27; First posted 2022-12-06 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections; Intra-Abdominal Infections; Skin and Soft Tissue Infection; Suspected Meningitis/Encephalitis or Any Other Infection; Sepsis
Keywords: Infection; mRNA; host response
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections; Intraabdominal Infections; Soft Tissue Infections; Encephalitis; Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NEWS2 score of 2-4: Bio-sample collection
  Interventions: Diagnostic Test: IMX-BVN-4 and IMX-SEV-4
- NEWS2 score of 5-6: Bio-sample collection
  Interventions: Diagnostic Test: IMX-BVN-4 and IMX-SEV-4
- NEWS2 score of ≥7: Bio-sample collection
  Interventions: Diagnostic Test: IMX-BVN-4 and IMX-SEV-4

INTERVENTIONS:
Diagnostic Test: IMX-BVN-4 and IMX-SEV-4 — Blood collection for mRNA analysis, Procalcitonin and CRP determination, molecular analysis of nasopharyngeal swab collection

SUMMARY:
This study aims to evaluate the diagnostic and prognostic performance of a novel mRNA diagnostic/prognostic classifier (interprets the expression of 29 host response mRNA biomarkers) from whole blood in adult patients presenting to emergency departments (ED) with suspected infection.

DETAILED DESCRIPTION:
Study measurements consists of a blood collection via venepuncture into a PAXgene® Blood RNA tube (2.5 ml) and Na-Heparin tube (4 ml) normally within 1 hour of enrolment into the study. The samples will be stored and transferred in batches from recruiting centres to a core laboratory. The expression of 29 mRNAs contained in the IMX-BVN-4/SEV-4 classifier will be analysed to determine the likelihood of bacterial and viral infection, as well as the likelihood of clinical deterioration. A nasopharyngeal swab sample will also be obtained for participants with suspected respiratory tract infection. Clinical data collection will be recorded from source data using an electronic Case Report Form (eCRF) The diagnosis of infection will be confirmed by a clinical adjudication panel blinded to the ED and hospital discharge diagnosis for each case.

ELIGIBILITY:
Inclusion Criteria:

Adult participants (16 years and older) presenting to the ED (or related assessment and treatment facilities such as SDEC or AMU) with:

1. Clinically suspected infection of any aetiology as the reason for attendance; AND
2. NEWS2 score of ≥2 (any dimension, using latest score)

Exclusion Criteria:

1. Treatment with systemic antibiotics, systemic antiviral agents or systemic antifungal agents within the past 7 days prior to the ED visit. Participants will not be excluded for use of:

   * Antiviral treatment for HIV infection and hepatitis B and hepatitis C
   * Topical antibiotics, topical antiviral or topical antifungal agents
   * Anti-herpes prophylaxis aiding suppression of a recuring herpes infection
   * Peri-operative (prophylactic) antibiotics
   * A single dose of antimicrobials during the present ED visit; note single dose can be considered mono- or combination therapy, wherein combination is administered as part of local Standard of Care and only one dose of each medication is administered
2. Presence of an advance directive to withhold life-sustaining treatment or a clear plan in place to that effect (ie. an explicit decision by patient/family/carer in conjunction with clinical team that active treatment beyond symptomatic relief is not appropriate). Note that patients who do not wish to receive cardiopulmonary resuscitation (CPR) but active treatment is still indicated may still qualify for entry into study
3. Prisoners or those in police custody
4. Patients who permanently lack the capacity to give informed consent
5. Previously enrolled in SPEED UK study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult participants (16 years and older) presenting to the ED (or related assessment and treatment facilities such as SDEC or AMU) with clinically suspected infection of any aetiology as the reason for attendance and a NEWS2 score of ≥2 (any dimension, using latest score)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1 | Admission
  Performance of the host response classifier IMX-BVN-4 to diagnose bacterial and viral infection as compared to clinical adjudication (sensitivity, specificity, likelihood ratios).
Primary Outcome 2 | Within 7 days after admission
  Prognostic performance of IMX-SEV-4 using an endpoint of receipt of critical-level care (including requirement for admission to critical care, mechanical ventilation, vasopressors (>12 hours), or renal replacement therapy) within 7 days (sensitivity, specificity, likelihood ratios).

SECONDARY OUTCOMES:
Secondary Outcome 1 | Up to 28 days after admission
  Prognostic performance of IMX-SEV-4 using a composite endpoint of Receipt of critical-level care (including requirement for transfer to critical care, mechanical ventilation, vasopressors (>12 hours), or renal replacement therapy) within 7 days, and/or 28-day in-hospital mortality (sensitivity, specificity, likelihood ratios).
Secondary Outcome 2 | Admission
  Diagnostic performance of the IMX-BVN-4 classifier in determining bacterial and viral infection compared with other biomarkers (procalcitonin and lactate) and clinical or laboratory findings obtained from standard of care, as compared to clinical adjudication (sensitivity, specificity, likelihood ratios).
Secondary Outcome 3 | Within 7 days after admission
  Prognostic performance of IMX-SEV-4 for clinical deterioration (NEWS2 of 5 or higher) within 7 days (sensitivity, specificity, likelihood ratios).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaieski DF, Mikkelsen ME, Band RA, Pines JM, Massone R, Furia FF, Shofer FS, Goyal M. Impact of time to antibiotics on survival in patients with severe sepsis or septic shock in whom early goal-directed therapy was initiated in the emergency department. Crit Care Med. 2010 Apr;38(4):1045-53. doi: 10.1097/CCM.0b013e3181cc4824. PMID 20048677
- [Background] Galtung N, Diehl-Wiesenecker E, Lehmann D, Markmann N, Bergstrom WH, Wacker J, Liesenfeld O, Mayhew M, Buturovic L, Luethy R, Sweeney TE, Tauber R, Kappert K, Somasundaram R, Bauer W. Prospective validation of a transcriptomic severity classifier among patients with suspected acute infection and sepsis in the emergency department. Eur J Emerg Med. 2022 Oct 1;29(5):357-365. doi: 10.1097/MEJ.0000000000000931. Epub 2022 Apr 21. PMID 35467566
- [Background] Bauer W, Kappert K, Galtung N, Lehmann D, Wacker J, Cheng HK, Liesenfeld O, Buturovic L, Luethy R, Sweeney TE, Tauber R, Somasundaram R. A Novel 29-Messenger RNA Host-Response Assay From Whole Blood Accurately Identifies Bacterial and Viral Infections in Patients Presenting to the Emergency Department With Suspected Infections: A Prospective Observational Study. Crit Care Med. 2021 Oct 1;49(10):1664-1673. doi: 10.1097/CCM.0000000000005119. PMID 34166284
- [Background] Brakenridge SC, Chen UI, Loftus T, Ungaro R, Dirain M, Kerr A, Zhong L, Bacher R, Starostik P, Ghita G, Midic U, Darden D, Fenner B, Wacker J, Efron PA, Liesenfeld O, Sweeney TE, Moldawer LL. Evaluation of a Multivalent Transcriptomic Metric for Diagnosing Surgical Sepsis and Estimating Mortality Among Critically Ill Patients. JAMA Netw Open. 2022 Jul 1;5(7):e2221520. doi: 10.1001/jamanetworkopen.2022.21520. PMID 35819783
- [Background] Brakenridge SC, Starostik P, Ghita G, Midic U, Darden D, Fenner B, Wacker J, Efron PA, Liesenfeld O, Sweeney TE, Moldawer LL. A Transcriptomic Severity Metric That Predicts Clinical Outcomes in Critically Ill Surgical Sepsis Patients. Crit Care Explor. 2021 Oct 14;3(10):e0554. doi: 10.1097/CCE.0000000000000554. eCollection 2021 Oct. PMID 34671746
- [Background] Sweeney TE, Shidham A, Wong HR, Khatri P. A comprehensive time-course-based multicohort analysis of sepsis and sterile inflammation reveals a robust diagnostic gene set. Sci Transl Med. 2015 May 13;7(287):287ra71. doi: 10.1126/scitranslmed.aaa5993. PMID 25972003
- [Background] Sweeney TE, Wong HR, Khatri P. Robust classification of bacterial and viral infections via integrated host gene expression diagnostics. Sci Transl Med. 2016 Jul 6;8(346):346ra91. doi: 10.1126/scitranslmed.aaf7165. PMID 27384347
- [Background] Sweeney TE, Perumal TM, Henao R, Nichols M, Howrylak JA, Choi AM, Bermejo-Martin JF, Almansa R, Tamayo E, Davenport EE, Burnham KL, Hinds CJ, Knight JC, Woods CW, Kingsmore SF, Ginsburg GS, Wong HR, Parnell GP, Tang B, Moldawer LL, Moore FE, Omberg L, Khatri P, Tsalik EL, Mangravite LM, Langley RJ. A community approach to mortality prediction in sepsis via gene expression analysis. Nat Commun. 2018 Feb 15;9(1):694. doi: 10.1038/s41467-018-03078-2. PMID 29449546
- [Background] Sweeney TE, Khatri P. Benchmarking Sepsis Gene Expression Diagnostics Using Public Data. Crit Care Med. 2017 Jan;45(1):1-10. doi: 10.1097/CCM.0000000000002021. PMID 27681387